CLINICAL TRIAL: NCT07364955
Title: Prospective Comparative Clinical Study of Three Parallel Cohorts on the Efficacy of Pre- and Post-surgical Vestibular Rehabilitation With or Without Rotary Stimulation in Patients With Vestibular Schwannoma
Brief Title: Vestibular Rehabilitation Protocol in Unilateral Vestibular Schwannoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Torrents Torrero (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Albert Torrents Torrero, Sub-Investigator Phd Student, Universitat Autonoma de Barcelona
Organization: Universitat Autonoma de Barcelona (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRV-SCHW25; PI-25-112 (Other: Research Ethics Committee oh Hospital Universitari Germans Trias i Pujol)
Record Dates: First submitted 2025-12-24; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Vestibular Schwannoma; Vestibular Schwannomas
Keywords: Vestibular rehabilitation; Vestibular prehabilitation; Vestibular prehab
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Intervention Model Description: Group 1) No-intervention group
  Group 2) Telerehabilitation program (ReHub) for 3 weeks before surgery and again for 3 weeks after surgery.
  Group 3) Rotatory Chair + Telerehabilitation program
Masking Description: Sequential convenience sampling approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM 1 - No Intervention Group (Other): Participants receive the standard surgical treatment for unilateral vestibular schwannoma and complete all study assessments (vHIT, DHI, posturography, hospital length of stay). They do not receive any pre- or postoperative vestibular rehabilitation.
  Interventions: Other: No Intervention: Observational Cohort
- ARM 2 - Group Telerehabilitation Only (Active Comparator): Participants complete a structured vestibular telerehabilitation program delivered through the ReHub digital platform for three weeks before surgery and for three weeks after surgery. The program includes guided home-based vestibular exercises, video instructions, activity tracking, and remote clinical supervision.
  Interventions: Behavioral: Structured home-based vestibular telerehabilitation program
- ARM 3 - Rotatory Chair + Telerehabilitation (Experimental): Participants receive the same vestibular telerehabilitation program as Arm 2 (three weeks before surgery and three weeks after surgery), plus six supervised preoperative sessions of controlled rotatory chair stimulation performed in the ENT department.
  Interventions: Behavioral: Structured home-based vestibular telerehabilitation program; Device: CE-marked clinical rotatory chair

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Participants undergo the standard surgical treatment for unilateral vestibular schwannoma and complete protocol assessments (vHIT, posturography, DHI, and hospital length of stay). They do not receive any preoperative or postoperative vestibular rehabilitation.
  Arms: ARM 1 - No Intervention Group
Behavioral: Structured home-based vestibular telerehabilitation program — Structured home-based vestibular rehabilitation program delivered through the ReHub digital platform for 3 weeks before surgery and 3 weeks after surgery, including gaze stabilization, balance, and habituation exercises with remote supervision.
  Arms: ARM 2 - Group Telerehabilitation Only; ARM 3 - Rotatory Chair + Telerehabilitation
Device: CE-marked clinical rotatory chair — Six supervised sessions of controlled vestibular stimulation delivered over 3 weeks using a CE-marked clinical rotatory chair following a progressive protocol in rotational velocity and post-rotation fixation tasks.
  Arms: ARM 3 - Rotatory Chair + Telerehabilitation

SUMMARY:
Brief Summary

The purpose of this clinical trial is to evaluate whether different strategies of vestibular rehabilitation, performed before and after surgery, can improve recovery in adults diagnosed with unilateral vestibular schwannoma. The main questions the study aims to answer are:

Does preoperative vestibular telerehabilitation improve postoperative vestibular compensation compared with no intervention?

Does adding preoperative rotatory chair stimulation to telerehabilitation lead to greater improvements in balance, dizziness, or hospital length of stay?

The study includes three comparison groups:

No-intervention group: Participants do not receive pre- or postoperative rehabilitation, but complete all study assessments (vHIT, DHI, posturography, and hospital length of stay).

Telerehabilitation group: Participants complete a structured home-based vestibular telerehabilitation program (ReHub) for 3 weeks before surgery and again for 3 weeks after surgery.

Rotatory Chair + Telerehabilitation group: Participants receive the same telerehabilitation program as the telerehabilitation group, plus six supervised sessions of preoperative rotatory chair stimulation (two sessions per week for three weeks), following a progressive protocol in the ENT department using a CE-marked clinical rotatory chair.

Participants will:

Attend routine preoperative and postoperative assessments (vHIT, posturography, and DHI).

Complete home-based vestibular exercises through a digital telerehabilitation platform (Groups 2 and 3).

If assigned to the Rotatory Chair + Telerehabilitation group, attend six in-hospital sessions of controlled rotatory chair stimulation during the three weeks before surgery.

Undergo follow-up evaluations at 4 and 12 weeks after surgery.

This study aims to determine whether structured vestibular training conducted before and after surgery can enhance postoperative compensation and reduce symptom burden in patients undergoing vestibular schwannoma surgery.

DETAILED DESCRIPTION:
This prospective, non-randomized, three-arm clinical trial evaluates the effect of two pre- and postoperative vestibular rehabilitation strategies on postoperative vestibular compensation in adults undergoing surgery for unilateral vestibular schwannoma. Aberrant vestibular compensation following vestibular neurectomy is common, and many patients experience prolonged imbalance, dizziness, altered gaze stabilization, and delayed return to functional independence. Early activation of vestibular adaptation, habituation, and substitution mechanisms may help optimize postoperative recovery.

The study compares three parallel cohorts:

a no-intervention group receiving standard clinical care,

a telerehabilitation group performing a structured home-based vestibular exercise program before and after surgery, and

an enhanced rehabilitation group receiving the same telerehabilitation program plus a progressive protocol of supervised preoperative rotatory chair stimulation.

Telerehabilitation is delivered through the ReHub platform, which provides guided vestibular exercises, real-time feedback, adherence tracking, and clinician monitoring. Preoperative rotatory stimulation consists of six supervised sessions over three weeks (two per week), following a structured progression in rotational velocity and post-rotation visual fixation tasks. The purpose of this stimulation is to facilitate preoperative habituation, improve gaze stabilization mechanisms, and prime central vestibular adaptation prior to the abrupt loss of vestibular function caused by surgery.

All participants undergo standardized assessments of vestibular function and balance control at predefined time points. These include the video Head Impulse Test (vHIT) to quantify VOR gain and refixation saccades, dynamic posturography to evaluate postural stability, and the Dizziness Handicap Inventory (DHI) to assess perceived disability. Hospital length of stay (LOS) is obtained directly from clinical records. Assessments are performed four weeks before surgery and at 4 and 12 weeks postoperatively.

The three-group design allows evaluation of:

1. the effect of pre- and postoperative vestibular telerehabilitation compared with no intervention,
2. the added effect of preoperative rotatory chair stimulation beyond telerehabilitation alone, and
3. the overall magnitude of combined preoperative rehabilitation strategies on functional recovery.

The study uses a sequential convenience sampling approach due to practical and ethical considerations related to implementation of the interventions. All data are collected at a tertiary referral center with specialized vestibular and neurotologic resources, ensuring standardized assessments and consistent clinical follow-up.

The primary objective is to compare postoperative vestibular compensation across groups, evaluated through changes in vHIT gain and refixation saccade patterns. Secondary objectives include differences in posturography metrics, DHI scores, and length of hospital stay. Additional exploratory analyses will examine the influence of age, sex, tumor size, and preoperative post-rotatory nystagmus inhibition time (TINPR) on rehabilitation outcomes.

The trial aims to generate evidence to inform future standardized rehabilitation pathways for patients undergoing vestibular schwannoma surgery, integrating digital rehabilitation tools and targeted vestibular stimulation to optimize central compensation mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Tumor size between 1.5 cm and 4 cm
* Unilateral vestibular schwannoma

Exclusion Criteria:

* Degenerative neurological conditions
* History of cerebrovascular disease
* Musculoskeletal deformities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Video Hit Impulse Test (VHIT) | Baseline (4 weeks before surgery), and at 3 and 12 weeks after surgery
posturography | Baseline (4 weeks before surgery), and at 3 and 12 weeks after surgery
Dizzines Handicap Inventory | Baseline (4 weeks before surgery), and at 3 and 12 weeks after surgery
  a 25-item self-reported questionnaire assessing perceived handicap due to dizziness, with total scores ranging from 0 to 100. Higher scores indicate greater perceived disability.
Lenght of hospital stay (LOS) | From surgery to hospital discharge (assessed at discharge)

SECONDARY OUTCOMES:
Post-rotatory nystagmus inhibition time (TINPR) | During each preoperative rotatory chair stimulation session (over the 3 weeks before surgery)
  only for group 3
Age | At enrollment
Sex | At enrollment
Tumor size | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified individual participant data underlying the results reported in publications arising from this study, including data related to primary and secondary outcomes such as vestibular function measures (e.g., vHIT parameters), posturography results, Dizziness Handicap Inventory (DHI) scores, and hospital length of stay. No directly identifiable personal data will be shared. Data will be available from 6 months after publication of the primary results and for up to 5 years thereafter, and will be shared with qualified researchers upon reasonable request and submission of a scientifically sound proposal related to vestibular rehabilitation or postoperative recovery. Approved data will be provided through secure institutional file transfer systems or controlled-access repositories, in accordance with applicable ethical approvals, informed consent, and data protection regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 6 months after publication of the primary study results and remaining available for 5 years thereafter.
Access Criteria: Access to de-identified individual participant data and supporting documentation will be granted to qualified researchers who submit a reasonable, methodologically sound research proposal related to vestibular rehabilitation, vestibular compensation, or postoperative recovery. Requests will be reviewed by the study investigators to ensure scientific merit, ethical compatibility, and alignment with the scope of the original study. Approved applicants will be required to agree to conditions of data use, including appropriate data protection measures and acknowledgment of the original study. Data will be shared through secure institutional file transfer systems or controlled-access repositories following approval.

REFERENCES:
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777
- [Background] Enticott JC, O'leary SJ, Briggs RJ. Effects of vestibulo-ocular reflex exercises on vestibular compensation after vestibular schwannoma surgery. Otol Neurotol. 2005 Mar;26(2):265-9. doi: 10.1097/00129492-200503000-00024. PMID 15793417
- [Background] Batuecas-Caletrio A, Santacruz-Ruiz S, Munoz-Herrera A, Perez-Fernandez N. The vestibulo-ocular reflex and subjective balance after vestibular schwannoma surgery. Laryngoscope. 2014 Jun;124(6):1431-5. doi: 10.1002/lary.24447. Epub 2013 Nov 13. PMID 24114593
- [Background] Gonzalez-Garcia M, Prieto-Sanchez-de-Puerta L, Montilla-Ibanez MA, Dominguez-Duran E, Sanchez-Gomez S, Sedeno-Vidal A. Efficacy of vestibular rehabilitation using unidirectional rotation paradigm in VOR asymmetry: systematic review and meta-analysis. Eur Arch Otorhinolaryngol. 2025 Aug;282(8):3845-3853. doi: 10.1007/s00405-025-09282-3. Epub 2025 Mar 18. PMID 40102225